CLINICAL TRIAL: NCT00178412
Title: Improving Outcomes of Hospitalized Elders and Caregivers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Bethel Powers, Principal Investigator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: R01NR008455-01 (NIH); R01NR008455 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Acute Illness
Keywords: Hospitalized elders; Family caregivers; Acute care
MeSH Terms: interventions — Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Treatment group
  Interventions: Behavioral: Care Project for Hospitalized Elders & Family Caregivers
- 2 (Active Comparator): Comparison Group
  Interventions: Behavioral: Comparison Group

INTERVENTIONS:
Behavioral: Care Project for Hospitalized Elders & Family Caregivers — Phase 1 in-hospital contact: Family caregivers complete baseline data, listen to a tape about helping the elderly relative cope with hospitalization, and work on a mutual agreement/identification of goals for participation in family member's hospital care (i.e., selection of two complications to focus on based on patient's illness condition)
  Phase 2 pre-hospital discharge: Family caregivers listen to a second tape about coping with the hospital experience, participating in their family member's in-hospital care, and preparing for hospital discharge/transition to home
  Arms: 1
Behavioral: Comparison Group — Phase 1 in-hospital contact: Family caregivers complete baseline data and listen to an informational tape about hospital policies.
  Phase 2 pre-hospital discharge: Family caregivers listen to a second informational tape about the hospital and medical center.
  Arms: 2

SUMMARY:
In this study, an intervention is tested that is designed to improve the outcomes of hospitalized elders and family caregivers.

Study design:

* randomized, controlled study
* participants: 280 family caregivers aged 21 or above
* length of follow-up: 2 weeks and 2 months after hospitalization

Study hypothesis: In this randomized clinical trial, the following hypotheses will be tested:

1. Hospitalized elders whose family CGs receive the CARE program versus those who receive a comparison program will have better outcomes during and after hospitalization as measured by: (1) fewer incidents of dysfunctional syndrome; (2) shorter hospital stays; (3) lower readmission rates; (4) less depressive symptoms; (5) higher cognitive level; (6) less functional decline perceived by family CG; and (7) a closer relationship with their family CGs.
2. Family CGs of hospitalized elders who receive the CARE program will report: (1) More positive beliefs about their loved one's responses to hospitalization and their role in the hospital setting; (2) more positive emotional outcomes (less worry, anxiety, and depressive symptoms) during and after hospitalization; (3) More participation in their loved one's care during hospitalization; and (4) More positive role outcomes (more role reward, less role strain, more prepared for their loved one's care, and a closer relationship with their elderly relatives, both during and after hospitalization).
3. The proposed model to explain the effects of the CARE program on the process and outcomes of family CG coping and elderly patient outcomes will be supported for CGs and elderly patients.

DETAILED DESCRIPTION:
More than 12 million elderly people are hospitalized each year in the United Status, frequently resulting in functional decline. Family care of hospitalized elders is important given the increasing numbers of hospitalized elders, needs for elder care in the home after hospital discharge, and responsibilities of family caregivers for providing this care. Involving family caregivers in the hospital care of their loved one may result in positive outcomes for both the elderly patients and their family caregivers. However, there is a paucity of empirical studies that have been conducted to evaluate the effectiveness of interventions to enhance family participation in caring for hospitalized elders. In the proposed study, we will build upon our prior work that has demonstrated the positive effects of theoretically-driven interventions with families of hospitalized patients and older adults at home. Among the unique contributions of this study include: (a) a randomized controlled design, (b) testing of a theoretically-driven, reproducible intervention that can be easily translated into clinical practice and widely disseminated; (c) the testing of an explanatory model to explain the effects of the intervention, (d) a prospective cost-effectiveness analysis; and (e) an intervention that begins early in the hospital stay, and (f) measurement of both short- and more long-term outcomes, up to 2 months following hospital discharge.

The primary aim of this study is to evaluate the effects of a theoretically-driven, reproducible intervention (CARE: Creating Avenues for Relative Empowerment) on the process and outcomes of hospitalized elders and their family caregivers. The secondary aims are to: (a) explore what factors moderate the effects of the intervention program (e.g., social economic status and family preferences for care participation); and (b) determine the cost-effectiveness of the CARE program. A two-group experiment will be used with 280 family caregivers of hospitalized elders. Measures of both process and outcome variables will be included, such as family caregiver beliefs, anxiety, worry, depression, role outcomes, as well as elderly patients outcomes during hospitalization and after hospital discharge. Findings from a recent pilot study with 49 family caregiver-elders dyads support undertaking this full-scale clinical trial in that family caregivers who received the CARE program, versus those who received a comparison program, had more positive coping and role outcomes and their hospitalized elderly relatives had positive outcomes during and after hospitalization.

ELIGIBILITY:
Inclusion Criteria:Family CGs

* age of 21 years or above;
* have an elderly relative (65 years or above) admitted to the three study units within the past 24-48 hours; (c) are related to the patient by blood, marriage, adoption, or affinity as a significant other (e.g., life partner, close friend);
* are primary CGs;
* can read and speak English; and
* live within a 1-hour drive of the facility (60 miles).

Exclusion Criteria: Family CGS

* paid care providers;
* unable to complete the questionnaires or provide care because of their own mental or physical impairment;

Patient:

* dies during the hospital stay or within 2 months after discharge;
* is transferred from the Intensive Care Unit (ICU) and stayed in the ICU for more than 2 nights;
* is diagnosed with dementia;
* is admitted from a long-term care facility; and
* is hospitalized for longer than 30 days
* is staying longer than 6 weeks in a nursing home immediately after hospitalization.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2003-04; Primary Completion 2006-04 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Patients' outcomes: rates of dysfunctional syndrome, readmission rate, and depression. | At intake, 1-3 days pre-hospital discharge, at 2 weeks and at 2 months post hospital discharge
Family Caregiver: emotional coping (worry, anxiety and depression); functional coping (participation in patient's care); and role outcomes(role reward, role strain) | 1-3 days pre-hospital discharge, at 2 weeks and at 2 months post hospital discharge

SECONDARY OUTCOMES:
Cost analysis. | At intake, 1-3 days pre-hospital discharge, at 2 weeks and at 2 months post hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Hong Li, Ph.D., RN, Principal Investigator — University of Rochester School of Nursing; Bethel A Powers, RN, PhD, Principal Investigator — University of Rochester School of Nursing
Locations (1):
- University of Rochester School of Nursing, Rochester, New York, United States

REFERENCES:
- [Background] Li H, Melnyk BM, McCann R. Review of intervention studies of families with hospitalized elderly relatives. J Nurs Scholarsh. 2004;36(1):54-9. doi: 10.1111/j.1547-5069.2004.04011.x. PMID 15098419
- [Background] Li H, Melnyk BM, McCann R, Chatcheydang J, Koulouglioti C, Nichols LW, Lee MD, Ghassemi A. Creating avenues for relative empowerment (CARE): a pilot test of an intervention to improve outcomes of hospitalized elders and family caregivers. Res Nurs Health. 2003 Aug;26(4):284-99. doi: 10.1002/nur.10091. PMID 12884417
- [Background] Li H. Family caregivers' preferences in caring for their hospitalized elderly relatives. Geriatr Nurs. 2002 Jul-Aug;23(4):204-7. doi: 10.1067/mgn.2002.126966. PMID 12183745
- [Result] Li H. Hospitalized elders and family caregivers: a typology of family worry. J Clin Nurs. 2005 Jan;14(1):3-8. doi: 10.1111/j.1365-2702.2004.01013.x. PMID 15656842
- [Result] Li H. Identifying family care process themes in caring for their hospitalized elders. Appl Nurs Res. 2005 May;18(2):97-101. doi: 10.1016/j.apnr.2004.06.015. PMID 15991107